CLINICAL TRIAL: NCT02380092
Title: A Multicentre, Prospective, Post Market Clinical Follow Up Study of the LEGION™ Primary Total Knee System With VERILAST™ Bearing Surface
Brief Title: Post Market Clinical Follow Up of LEGION™ Primary TKS With VERILAST™
Status: Active, not recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 12-4042-01
Record Dates: First submitted 2015-02-27; First posted 2015-03-05 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Joint Disease
Keywords: Knee; Post-Market Surveillance; Legion; Verilast; Degenerative Joint Disease
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LEGION™ Primary TKS with VERILAST™ Bearing Surface — All study subjects will be treated with LEGION™ Primary TKS with VERILAST™ Bearing Surface as per standard clinical practice.

SUMMARY:
LEGION™ Primary Total Knee System is CE-marked and marketed in all study regions. This study serves as post-market surveillance for LEGION™ Primary Total Knee System with the VERILAST™ bearing surface (OXINIUM™ femoral component with highly cross-linked polyethylene tibial insert).

All study subjects will receive a LEGION™ Primary Total Knee System with VERILAST™ bearing surface and the results will be analysed against historical data from patients who received a Genesis II knee replacement.

DETAILED DESCRIPTION:
The LEGION™ Primary Total Knee System (TKS) is a comprehensive, state-of-the-art system that empowers surgeons to address diverse surgical challenges and provide personalized joint care. The LEGION™ Primary TKS implant designs were built on the legacy of the GENESIS™ II TKS. For more than 15 years and in more than 30 countries, the GENESIS™ II TKS has achieved outstanding clinical outcomes.

As CE-mark and 510k approval for the LEGION™ Primary TKS has been obtained, it is being used in clinical practice in several countries including Europe and the US but clinical studies need to be carried out in order to confirm its safety and efficacy and in order to conform to the medical device directives (MEDDEV. 2.7.1 Rev.3).

This study is therefore a post-market study to evaluate the short-, mid- and long-term safety and effectiveness of the LEGION™ Primary TKS with VERILAST™ bearing surface (the combination of an OXINIUM™ femoral component with highly cross-linked polyethylene tibial base plate inserts). The clinical outcome from a large cohort of subjects who are treated with the LEGION™ Primary TKS as part of their standard of care will be documented. The study is designed to reflect standard clinical practice as closely as possible because it allows the results of such a study to represent the true clinical outcome that would be achieved in clinical practice, up to a maximum. Only subjects who will be treated with the LEGION™ Primary TKS as part of their normally planned care will screened for participation in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires primary TKA and has elected to use the LEGION™ Primary TKS with VERILAST™.
* Subject requires primary TKA due to degenerative joint disease (primary osteoarthritis, post-traumatic arthritis, avascular necrosis, rheumatoid arthritis).
* Subject is of legal age to consent, agrees to consent to and to follow the study visit schedule (as defined in the study protocol and informed consent form), by signing the EC approved informed consent form.
* Routine radiographic assessment is possible.
* Subject plans to be available through ten (10) years postoperative follow-up.
* Subject is 18-75 years of age at the time of surgery.

Exclusion Criteria:

* Age > 75 years at the time of surgery.
* Subjects with immunosuppressive disorders.
* Subject has severe pronation of the ipsilateral foot or any other relevant clinical condition contributing to abnormal ambulation (including but not limited to ankle fusion, ankle arthroplasty, previous hip fracture, ipsilateral hip arthritis resulting in flexion contracture).
* Subject has undergone a previous major surgery to the study knee (including osteotomy, fracture fix, medial or lateral ligament surgery).
* Subject has active infection or sepsis (treated or untreated).
* At the time of enrollment, subject has one or more of the following arthroplasties that are not fully healed and well-functioning, as determined by the Investigator:

  * Ipsilateral or contralateral primary total hip arthroplasty or hip resurfacing arthroplasty.
  * Contralateral primary total knee or unicondylar knee arthroplasty.
* Subject has presence of malignant tumor, metastatic, or neoplastic disease.
* Subject has conditions that may interfere with the TKA survival or outcome (i.e., Paget's or Charcot's disease, muscular atrophy, uncontrolled diabetes, moderate to severe renal insufficiency or neuromuscular disease).
* Subject has any acute or chronic morbidity of vascular origin that, in the opinion of the Investigator, is likely to compromise successful treatment or compliance to follow-up visits.
* Subject has inadequate bone stock to support the device (severe osteopenia, family history of severe osteoporosis or osteopenia).
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study.
* Subject has a Body Mass Index (BMI) >40.0.
* Subject requires revision TKA.
* Subject is expected to require bilateral TKA within 1 year following study knee replacement.
* Subject does not understand the language used in the Informed Consent Form.
* Subject is enrolled in another clinical study at the same time.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are scheduled to have Total Knee Arthroplasty with the Legion Primary Total Knee System due to Degenerative Joint Disease.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Survival | 10 years
  Non-inferiority of survival of Legion Primary with Verilast compared to a literature reference rate of 92.6% for Genesis II TKS

SECONDARY OUTCOMES:
Number of revisions | Discharge, 3 months, 1 year, 3 years, 5 years, 7 years, 10 years
  Number of revisions (of any component of the device) at all follow up timepoints
Changes in mean 2011 Knee Society Score | Discharge, 3 months, 1 year, 3 years, 5 years, 10 years
  Changes in mean 2011 Knee Society Score from baseline to each subsequent assessment
Changes in mean Euroqol 5-D score | Discharge, 3 months, 1 year, 3 years, 5 years, 10 years
  Changes in mean Euroqol 5-D score from baseline to each subsequent assessment
Changes in radiographic evaluation | Discharge, 3 months, 1 year, 3 years, 5 years, 10 years
  Changes in radiographic evaluation from baseline to each subsequent assessment
AEs | Operative, Discharge, 3 months, 1 year, 3 years, 5 years, 7 years, 10 years
  Adverse Event reporting from surgery to 10 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Karlie Morgan, Study Director — Director of Clinical Study Management, Global Clinical Research Operations
Locations (7):
- Austria (2):
  - Evangelisches Krankenhaus Wien, Vienna
  - Orthopadische Krankenhaus Gersthof, Vienna
- Germany (4):
  - AMEOS Klinikum Seepark Geestland, Langen, Kreis Geestland
  - OrthoCentrum, Hamburg
  - CaritasKlinikum St. Joseph Saarbrücken-Dudweiler, Saarbrücken-Dudweiler
  - KniePraxis Prof. Dr. Tibesku, Straubing
- Servicio de C.O.T. Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Spain